CLINICAL TRIAL: NCT03057548
Title: Left Atrial Posterior Wall Isolation in Conjunction With Pulmonary Vein Isolation for Treatment of Persistent Atrial Fibrillation (PIVoTAL) Trial
Brief Title: Comparison of Pulmonary Vein Ablation With or Without Left Atrial Posterior Wall Ablation for Persistent AF (PIVoTAL)
Acronym: PIVoTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arash Aryana, MD (Other)
Responsible Party: Sponsor-Investigator, Arash Aryana, MD, Cardiac Electrophysiologist / Principal Investigator, Sacramento EP Research
Organization: Sacramento EP Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIVotal-01
Record Dates: First submitted 2017-02-08; First posted 2017-02-20 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation Chronic; Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Long-Standing Atrial Fibrillation; Posterior Left Atrial Wall Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Vein Isolation (PVI) (Active Comparator): Cryoablation only of Pulmonary Veins
  or
  Radiofrequency ablation only of Pulmonary Veins
  Pulmonary Vein Isolation (PVI) alone.
  Interventions: Procedure: Cryo or Radiofrequency (RF) Ablation only of Pulmonary Veins
- PVI & Posterior Left Atrial Ablation (Experimental): Cryoablation of Pulmonary Veins plus RF ablation of Posterior Left Atrial Wall
  or
  Radiofrequency ablation of Pulmonary Veins plus RF ablation of Posterior Left Atrial Wall
  PVI ablation plus ablation of the Posterior Left Atrial Wall (PLAW)
  Interventions: Procedure: Cryo or RF Ablation of Pulmonary Veins plus Ablation of the PLAW

INTERVENTIONS:
Procedure: Cryo or Radiofrequency (RF) Ablation only of Pulmonary Veins — Artic Front Advance Cardiac Cryoablation System used to ablate the Pulmonary Veins
  OR
  FDA Approved RF Ablation Catheter used to ablate the Pulmonary Veins.
  Ablation of the Pulmonary Veins alone
  Other Names: Artic Front Advance Cardiac Cryoablation System; FDA Approved Radiofrequency Ablation Catheter
  Arms: Pulmonary Vein Isolation (PVI)
Procedure: Cryo or RF Ablation of Pulmonary Veins plus Ablation of the PLAW — Cryoablation of the Pulmonary Veins plus RF Ablation of the PLAW
  OR
  RF Ablation of the Pulmonary Veins plus RF Ablation of the PLAW
  Ablation of the Pulmonary Veins plus RF ablation of the Posterior Left Atrial Wall (PLAW)
  Other Names: Cryoablation of Pulmonary Veins plus RF Ablation of PLAW; RF Ablation of Pulmonary Veins plus RF Ablation of PLAW
  Arms: PVI & Posterior Left Atrial Ablation

SUMMARY:
The purpose of this study it to learn whether pulmonary vein isolation (PVI) along with ablation of the posterior left atrial wall (PLAW) will reduce the likelihood of atrial fibrillation (AF) recurrence in patients with persistent or long-standing persistent AF one year after an ablation procedure in comparison to a PVI ablation procedure, alone.

The investigator hypothesizes that the combination of PVI plus PLAW isolation will result in a reduction in recurrence of atrial arrhythmias at one year after ablation.

DETAILED DESCRIPTION:
Patients with persistent or long-standing persistent atrial fibrillation will be enrolled in this multi-center, randomized, prospective, single-blinded study. All patients are required to be in atrial fibrillation (AF) on the day of the ablation procedure. After ablation (isolation) of the pulmonary veins (PVI) is complete, and while still in the electrophysiology lab, all patients are randomized to either PVI, alone [Group 1] or the combination of PVI plus ablation of the posterior left atrial wall (PLAW) [Group 2]. For those patients randomized to PVI, their ablation procedure is complete at this time. For those patients randomized to PVI plus PLAW, they will have the additional ablation to the posterior left atrial wall performed.

All study patients have the same follow-up after their ablation procedure: clinic visits at 3, 6, and 13 months; a heart event monitor is worn for 7-14 days before these visits. An echocardiogram is done at 4-6 months after the ablation procedure. Blood thinners are usually recommended for three months after the ablation procedure and then the need for continued use of blood thinners will be based on individual patient's medical history, stroke risk and the judgement of their study doctor. Information about patient's medical history, heart arrhythmias, and atrial fibrillation will be collected during the study. This information will be analyzed as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with an age >18 years undergoing a first-time catheter ablation of AF; prior ablation of a right atrial cardiac arrhythmia (i.e., typical right atrial flutter) is permitted
* All patients must understand the requirements of the study and be willing to comply with the post-study follow-up requirements
* Patients must be in AF on the day of the procedure

Exclusion Criteria:

* Any reversible cause of AF (post-operative, thyroid disorder, etc)
* Patients with cerebral ischemic events (stroke or transient ischemic attack), myocardial infarction or unstable angina in the previous 2 months
* Patients with any corrected or uncorrected congenital heart disease
* Patients with a history of hypertrophic cardiomyopathy
* Patients with cardiomyopathy and a left ventricular ejection fraction <35%
* Congestive heart failure, class IV
* Women who are known to be pregnant or have had a positive β-Human Chorionic Gonadotropin (β-HCG) test 7 days prior to procedure
* Patients whose life expectancy is <1 year
* History of left-sided left atrial ablation (catheter or surgically-based)
* Mental impairment precluding the patient from providing informed consent or completing appropriate follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arash Aryana, MD, Principal Investigator — Mercy General Hospital and Dignity Health Heart and Vascular Institute
Locations (2):
- Mercy General Hospital and Dignity Health Heart and Vascular Institute, Sacramento, California, United States
- Heart Center, Japan Red Cross Yokohama-city Bay Hospital, Yokohama, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Brooks AG, Stiles MK, Laborderie J, Lau DH, Kuklik P, Shipp NJ, Hsu LF, Sanders P. Outcomes of long-standing persistent atrial fibrillation ablation: a systematic review. Heart Rhythm. 2010 Jun;7(6):835-46. doi: 10.1016/j.hrthm.2010.01.017. Epub 2010 Jan 22. PMID 20206320
- [Background] Segerson NM, Daccarett M, Badger TJ, Shabaan A, Akoum N, Fish EN, Rao S, Burgon NS, Adjei-Poku Y, Kholmovski E, Vijayakumar S, DiBella EV, MacLeod RS, Marrouche NF. Magnetic resonance imaging-confirmed ablative debulking of the left atrial posterior wall and septum for treatment of persistent atrial fibrillation: rationale and initial experience. J Cardiovasc Electrophysiol. 2010 Feb;21(2):126-32. doi: 10.1111/j.1540-8167.2009.01611.x. Epub 2009 Oct 5. PMID 19804549
- [Background] Cutler MJ, Johnson J, Abozguia K, Rowan S, Lewis W, Costantini O, Natale A, Ziv O. Impact of Voltage Mapping to Guide Whether to Perform Ablation of the Posterior Wall in Patients With Persistent Atrial Fibrillation. J Cardiovasc Electrophysiol. 2016 Jan;27(1):13-21. doi: 10.1111/jce.12830. Epub 2015 Oct 30. PMID 26515166
- [Background] Elbatran AI, Anderson RH, Mori S, Saba MM. The rationale for isolation of the left atrial pulmonary venous component to control atrial fibrillation: A review article. Heart Rhythm. 2019 Sep;16(9):1392-1398. doi: 10.1016/j.hrthm.2019.03.012. Epub 2019 Mar 16. PMID 30885736
- [Background] Corradi D, Callegari S, Maestri R, Ferrara D, Mangieri D, Alinovi R, Mozzoni P, Pinelli S, Goldoni M, Privitera YA, Bartoli V, Astorri E, Macchi E, Vaglio A, Benussi S, Alfieri O. Differential structural remodeling of the left-atrial posterior wall in patients affected by mitral regurgitation with or without persistent atrial fibrillation: a morphological and molecular study. J Cardiovasc Electrophysiol. 2012 Mar;23(3):271-9. doi: 10.1111/j.1540-8167.2011.02187.x. Epub 2011 Sep 28. PMID 21954878
- [Background] Nagashima K, Okumura Y, Watanabe I, Nakahara S, Hori Y, Iso K, Watanabe R, Arai M, Wakamatsu Y, Kurokawa S, Mano H, Nakai T, Ohkubo K, Hirayama A. Hot Balloon Versus Cryoballoon Ablation for Atrial Fibrillation: Lesion Characteristics and Middle-Term Outcomes. Circ Arrhythm Electrophysiol. 2018 May;11(5):e005861. doi: 10.1161/CIRCEP.117.005861. PMID 29700055
- [Background] Okumura Y, Watanabe I, Iso K, Takahashi K, Nagashima K, Sonoda K, Mano H, Yamaguchi N, Kogawa R, Watanabe R, Arai M, Ohkubo K, Kurokawa S, Nakai T, Hirayama A. Mechanistic Insights Into Durable Pulmonary Vein Isolation Achieved by Second-Generation Cryoballoon Ablation. J Atr Fibrillation. 2017 Apr 30;9(6):1538. doi: 10.4022/jafib.1538. eCollection 2017 Apr-May. PMID 29250289
- [Background] Reddy VY, Sediva L, Petru J, Skoda J, Chovanec M, Chitovova Z, Di Stefano P, Rubin E, Dukkipati S, Neuzil P. Durability of Pulmonary Vein Isolation with Cryoballoon Ablation: Results from the Sustained PV Isolation with Arctic Front Advance (SUPIR) Study. J Cardiovasc Electrophysiol. 2015 May;26(5):493-500. doi: 10.1111/jce.12626. Epub 2015 Apr 15. PMID 25644659
- [Background] Aryana A, Baker JH, Espinosa Ginic MA, Pujara DK, Bowers MR, O'Neill PG, Ellenbogen KA, Di Biase L, d'Avila A, Natale A. Posterior wall isolation using the cryoballoon in conjunction with pulmonary vein ablation is superior to pulmonary vein isolation alone in patients with persistent atrial fibrillation: A multicenter experience. Heart Rhythm. 2018 Aug;15(8):1121-1129. doi: 10.1016/j.hrthm.2018.05.014. PMID 30060879
- [Background] Nishimura T, Yamauchi Y, Aoyagi H, Tsuchiya Y, Shigeta T, Nakamura R, Yamashita M, Asano M, Nakamura T, Suzuki H, Shimura T, Kurabayashi M, Keida T, Sasano T, Hirao K, Okishige K. The clinical impact of the left atrial posterior wall lesion formation by the cryoballoon application for persistent atrial fibrillation: Feasibility and clinical implications. J Cardiovasc Electrophysiol. 2019 Jun;30(6):805-814. doi: 10.1111/jce.13879. Epub 2019 Feb 23. PMID 30767365
- [Background] Aryana A, Kenigsberg DN, Kowalski M, Koo CH, Lim HW, O'Neill PG, Bowers MR, Hokanson RB, Ellenbogen KA; Cryo-DOSING Investigators. Verification of a novel atrial fibrillation cryoablation dosing algorithm guided by time-to-pulmonary vein isolation: Results from the Cryo-DOSING Study (Cryoballoon-ablation DOSING Based on the Assessment of Time-to-Effect and Pulmonary Vein Isolation Guidance). Heart Rhythm. 2017 Sep;14(9):1319-1325. doi: 10.1016/j.hrthm.2017.06.020. Epub 2017 Jun 15. PMID 28625929
- [Background] Markides V, Schilling RJ, Ho SY, Chow AW, Davies DW, Peters NS. Characterization of left atrial activation in the intact human heart. Circulation. 2003 Feb 11;107(5):733-9. doi: 10.1161/01.cir.0000048140.31785.02. PMID 12578877

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulmonary Vein Isolation (PVI): Cryoablation only of Pulmonary Veins
  or
  Radiofrequency (RF) ablation only of Pulmonary Veins
  Pulmonary Vein Isolation (PVI) alone.
  Cryo or RF Ablation only of Pulmonary Veins: Artic Front Advance Cardiac Cryoablation System used to ablate the Pulmonary Veins
  OR
  FDA Approved RF Ablation Catheter used to ablate the Pulmonary Veins.
  Ablation of the Pulmonary Veins alone
- PVI & Posterior Left Atrial Ablation: Cryoablation of Pulmonary Veins plus RF ablation of Posterior Left Atrial Wall
  or
  Radiofrequency ablation of Pulmonary Veins plus RF ablation of Posterior Left Atrial Wall
  PVI ablation plus ablation of the Posterior Left Atrial Wall (PLAW)
  Cryo or RF Ablation of Pulmonary Veins plus Ablation of the PLAW: Cryoablation of the Pulmonary Veins plus RF Ablation of the PLAW
  OR
  RF Ablation of the Pulmonary Veins plus RF Ablation of the PLAW
  Ablation of the Pulmonary Veins plus RF ablation of the Posterior Left Atrial Wall (PLAW)
Period: Overall Study
Arm/Group | Pulmonary Vein Isolation (PVI) | PVI & Posterior Left Atrial Ablation
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pulmonary Vein Isolation (PVI): Cryoablation only of Pulmonary Veins
  or
  Radiofrequency ablation only of Pulmonary Veins
  Pulmonary Vein Isolation (PVI) alone.
  Cryo or RF Ablation only of Pulmonary Veins: Artic Front Advance Cardiac Cryoablation System used to ablate the Pulmonary Veins
  OR
  FDA Approved RF Ablation Catheter used to ablate the Pulmonary Veins.
  Ablation of the Pulmonary Veins alone
- Total: Total of all reporting groups
Arm/Group | Pulmonary Vein Isolation (PVI) | PVI & Posterior Left Atrial Ablation | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 26 | 46
  >=65 years | 35 | 29 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9) | 67 (8) | 68.5 (2.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 33 | 35 | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 21 | 47
  Japan | 29 | 34 | 63
Long-standing persistent atrial fibrillation [Count of Participants; unit: Participants] | 17 | 21 | 38
Persistent atrial fibrillation [Count of Participants; unit: Participants] | 38 | 34 | 72

OUTCOME MEASURES:

1. Primary Outcome: 1-year Freedom From Recurrent Atrial Arrhythmias
Description: The results of 7-14 day ambulatory ECG monitoring and ECGs performed at 3, 6 and 12 months will be used to document freedom from recurrent atrial fibrillation at one year post-ablation.
Time Frame: One year
Population: Study cohort consisted of patients undergoing first-time cryoballoon ablation for symptomatic persistent/long-standing persistent atrial ablation (55 subjects in the PVI isolation arm and 55 subjects in the PVI+PWI arm) were analyzed for freedom from recurrence of atrial fibrillation and all atrial arrhythmias at one-year post-study ablation.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulmonary Vein Isolation (PVI) | PVI & Posterior Left Atrial Ablation
Number analyzed (Participants) | 55 | 55
Participants | 25 | 14

2. Secondary Outcome: Overall Complication Rate
Description: The type and frequency of complications following catheter ablation
Time Frame: During follow-up, assessed for an estimated total of one year.
Measure: Count of Participants; unit: Participants
Groups:
- Pulmonary Vein Isolation (PVI): Cryoablation only of Pulmonary Veins
  or
  Radiofrequency ablation only of Pulmonary Veins
  Pulmonary Vein Isolation (PVI) alone.
  Cryo or Radiofrequency (RF) Ablation only of Pulmonary Veins: Artic Front Advance Cardiac Cryoablation System used to ablate the Pulmonary Veins
  OR
  FDA Approved RF Ablation Catheter used to ablate the Pulmonary Veins.
  Ablation of the Pulmonary Veins alone
Arm/Group | Pulmonary Vein Isolation (PVI) | PVI & Posterior Left Atrial Ablation
Number analyzed (Participants) | 55 | 55
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 1 year following the study ablation procedure.
Description: All study subjects were queried regarding any adverse or serious adverse events at each study visit (3, 6 and 12 months post-study ablation procedure). Additionally, the investigator and research coordinator reviewed each subject's electronic medical record at the time of all study visits to assess for any adverse events not reported by the subjects.
Groups:
- PVI Only: The incidence of adverse events was 5.5% in PVI only group.
- PVI+PWI: The incidence of adverse events was 5.5% in PVI+PWI group.
Arm/Group | PVI Only | PVI+PWI
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 3/55 | 3/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PVI Only (N=55) | PVI+PWI (N=55)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0) — Congestive Heart Failure Exacerbation
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Persistent Phrenic Nerve Palsy (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Symptomatic bradycardia requiring implantation of a permanent pacemaker
Groin Vascular Complication (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Slight variations in ablation strategy/periprocedural management may have existed among operators. Baseline Left Atrial Posterior Wall low-voltage data were collected in AF at procedure start, which could have implications. Subclinical manifestations of complications (ex. esophageal ulcerations or asymptomatic PV stenosis) could not be excluded as diagnostic studies weren't performed in follow-up. Recurrent asymptomatic atrial arrhythmias could have occurred without detection during follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT03057548/Prot_000.pdf
  • Informed Consent Form (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT03057548/ICF_001.pdf